CLINICAL TRIAL: NCT01294111
Title: Tai Chi Training for Elderly People With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Stiftelsen Ronnbaret (Unknown); The Swedish Heart and Lung Association (Other); Visare Norr (Unknown)
Responsible Party: Principal Investigator, Lena Hagglund, RNT, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tai Chi for heart failure
Record Dates: First submitted 2011-01-03; First posted 2011-02-11 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Chronic Heart Failure
Keywords: Fatigue; Quality of life; Elderly
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Tai Chi training (Experimental): Participation in a group of 15 patients, completing a 60 minutes tai chi training programme twice-weekly for 16 weeks.
  Interventions: Behavioral: Tai Chi training
- Control (No Intervention): Living as usual, following ordinary care plans and personal activities. Participants will be called to hospital for data collection. Participants are asked not to start any of the activities Tai Chi, Qui Gong or Yoga during the study period.

INTERVENTIONS:
Behavioral: Tai Chi training — Three groups with 15 participants each will complete a 60 minutes tai chi training programme twice-weekly for 16 weeks. The programme is worked out by an expert in Chinese traditional medicine to suit elderly people with chronic heart failure, and the classes are led by experienced leaders.
  Arms: Tai Chi training

SUMMARY:
Physical activity is recommended in the treatment of heart failure. Elderly people demand various forms of physical activity. Tai chi has shown to be an appreciated form of physical activity among elderly, although there is a lack of studies focusing people aged 70 years and older.

The overall goal with the project is to find a form of physical activity that is safe and free from side effects, suitable for elderly people with chronic heart failure. The hypothesis is that for patients participating in tai chi training during three months the degree of self rated fatigue will be reduced and health-related quality of life will increase, compared with a control group receiving ordinary care. The primary aim is to study the effect of tai chi training on fatigue and health-related quality of life. A second aim is to study effects on physical function and levels of brain natriuretic peptide (BNP) in blood plasma. A tertiary aim is to describe the experience of participating in tai chi training.

A mixed methods study is conducted. Fortyfive patients with a verified diagnosis of heart failure in the age of 70 years or older, who experience fatigue according to the Multi Fatigue Inventory (MFI-20), was randomized to intervention or control group. Three groups with 8-9 participants each completed a tai chi training programme twice-weekly for 16 weeks. Data was collected at baseline, directly after the 16 weeks of training, and 6 and 12 months thereafter. The programme is worked out by an expert in Chinese traditional medicine to suit elderly people with chronic heart failure, and the classes were led by experienced leaders. Before the start of the study a small pilot study was conducted to test the feasibility of the programme. A group of seven patients completed the programme for eight weeks without any problems.

If tai chi has a good effect on fatigue, health-related quality of life and physical function, this form of physical activity can be a valuable complement to other medical treatment. Tai chi has a potential to be offered to many patients to a relatively low cost. It can be practiced in groups or in private, and also through internet connection.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of heart failure
* Left ventricle ejection fraction < 50
* Stable medical treatment with Angiotensin Converting Enzyme blockers and Betareceptor blockers (if no contraindications) experience of fatigue according to the Multidimensional Fatigue Inventory
* 70 years or older
* Swedish speaking

Exclusion Criteria:

* Instable angina pectoris
* Myocardial infarction within the last three months
* Cognitive impairment
* No experienced fatigue

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline values of the Multidimensional Fatigue Inventory, MFI-20 | after intervention of 16 weeks, at 6 months and 12 months after intervention
  A self-report instrument of five dimensions of fatigue. General fatigue, physical fatigue, mental fatigue, reduced activity and reduced motivation.

SECONDARY OUTCOMES:
Changes from baseline values of the Minnesota Living With Heart Failure Questionnaire (LHFQ) | after intervention of 16 weeks, at 6 months and 12 months after intervention
  A self-report instrument aimed to measure the effects of symptoms, functional limitations and psychological distress on an individual´s quality of life.

OTHER OUTCOMES:
To describe the experience of participating in tai chi training | after completed intervention
  Qualitative individual interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Umea University, Skellefteå, Västerbotten County, Sweden

REFERENCES:
- [Background] Barrow DE, Bedford A, Ives G, O´Toole LO, & Channer KS (2007). An evaluation of the effects of Tai Chi Chuan and Chi Kung training in patients with symptomatic heart failure: a randomised controlled pilot study. Postgrad Med, 83,717-721. Cheng TO (2007). Tai Chi: The Chinese ancient wisdom of an ideal exercise for cardiac patients. Int J Cardiol, 117, 293-295. (editorial) Dolansky MA, Moore SM, & Visovsky C (2006). Older adults´ views of cardiac rehabilitation programs. J Gerontol Nurs, 32(2), 37-44. Hägglund, L., Boman, K., Stenlund, H., Lundman, B., & Brulin, C. (2008). Factors related to fatigue among older patients with heart failure in primary health care. Int J Older People Nurs, 3(2), 96-103. Motivala SJ, Sollers J, Thayer J & Irwin MR (2006). Tai Chi Chih acutely decreases sympathetic nervous system activity in older adults. J Ger A Bio Sci Med, 61(11), 1177-1180. Rector TS, Kubo SH, & Cohn JN (1987). Patients´self-assessment of their congestive heart failure: Part 2: Content, reliability and validity of a new measure, The Minnesota Living with Heart Failure Questionnaire. Heart Fail, 3, 198-209. Rees K, Taylor RS, Singh S, Coats AJS, & Ebrahim S (2004). Exercise based rehabilitation for heart failure. Cochrane Database of Systematic Reviews, (3) Art.No.: CD003331. DOI: 10.1002/14651858.CD003331.pub2. Smets EMA, Garssen B, Bonke B, de Haes JCJM. 1995. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res, 39 (5), 315-25. Verhagen AP, Immink M, van der Meulen A, & Bierma-Zeinstra SMA (2004). The efficacy of Tai Chi Chuan in older adults: a systematic review. Fam Pract, 21, 107-113. Yeh GY, Wood MJ, Lorell BH, Stevenson LW, Eisenberg DM, Wayne PM, Goldberger AL, Davis RB, & Phillips RS. (2004). Effects of Tai Chi mind-body movement therapy on functional status and exercise capacity in patients with chronic heart failure: A randomized controlled trial. Am J Med, 117, 541-548.